CLINICAL TRIAL: NCT03556917
Title: The Effects of Iontophoresis in Women With Gynoid Hidrolipodystrophy.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universidade Norte do Paraná (Other)
Responsible Party: Principal Investigator, Alana Roberta Quessada, Master student, Universidade Norte do Paraná
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2.264.773
Record Dates: First submitted 2018-05-15; First posted 2018-06-14 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Caffeine; Cellulitis
MeSH Terms: conditions — Cellulitis | interventions — Iontophoresis; Caffeine

STUDY DESIGN:
Intervention Model Description: It is a longitudinal and randomized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- group 1 (Active Comparator): topical gel base + caffeine.
  Interventions: Combination Product: iontophoresis + caffeine
- group 2 (Active Comparator): iontophoresis + caffeine
  Interventions: Combination Product: iontophoresis + caffeine
- Group 3 (Active Comparator): iontophoresis
  Interventions: Combination Product: iontophoresis + caffeine

INTERVENTIONS:
Combination Product: iontophoresis + caffeine — we will use cafeislaine c (caffeine) +galvanic current

SUMMARY:
Introduction: Gynoid hydrolipodystrophy (HLDG) or cellulitis is a subcutaneous tissue disorder, with several strategies for its treatment, such as caffeine and iontophoresis. Objective: To evaluate the effects of caffeine-associated iontophoresis for the treatment of HLDG. Methods: In a longitudinal study, participants will be evaluated for: photographic documentation, ultrasound imaging, thermography and quality of life questionnaire. If included, they will be separated into 3 randomized groups (n = 30). G1: use of base gel (n = 10); G2: use of iontophoresis and gel with caffeine (n = 10) and G3: use of iontophoresis alone (n = 10). The groups will be treated with 10 sessions, 2 times per week. After that they will be reevaluated. Statistical analysis: The software used will be the SPSS StatisticalPackage (IBM SPSS Statistics, Chicago, IL, USA). The data distribution will be analyzed by the Shapiro-Wilk test. In case of normal distribution, the data will be described as mean ± standard deviation; otherwise, as median [interquartile range 25-75%]. For comparison of the data, we will use ANOVA and for comparison of means the Tukey test and case not normal distribution, krulskal-Wallis test and the Dunns test. The level of statistical significance adopted will be P <0.05. Expected contributions: It is expected that investigators can contribute to the treatment of patients with HLDG and analyze the effects of iontophoresis with caffeine, both in clinical and scientific practice, providing a method that is valid and reliable for this purpose; multidisciplinary training of highly qualified human resources and the strengthening and consolidation of a research team.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild to moderate cellulite diagnosis will be included, according to the validated Photonumeric scale of cellulite severity
* Body mass index less than 30 (kg / m2)

Exclusion Criteria:

* Individuals who have a deregulated menstrual cycle who are pregnant;
* Breastfeeding or using some hormone;
* Antibiotic medication including steroids over 1 month of treatment of skin diseases; •Sensitivity or hypersensitivity of the skin;
* Use of the same or similar cosmetics or remedies on the glutes within 1 month;
* Surgical procedure (liposuction and skin treatments) in the region to be treated or planning some procedure within the study period;
* Chronic debilitating diseases such as asthma, diabetes or hypertension;
* Atopic dermatitis

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-06-14 (Actual); Primary Completion 2019-03-17 (Actual); Study Completion 2019-04-04 (Actual)

PRIMARY OUTCOMES:
thickness | through study completion, an average of 1 year.
  change from baseline subcutaneous adipose tissue thickness at after 10 sessions

SECONDARY OUTCOMES:
temperature | through study completion, an average of 1 year.
  change from baseline superficial temperature of the gluteous skin at after 10 sessions
score quality of life | through study completion, an average of 1 year.
  change from baseline quality of life impact in patients with cellulits at after 10 sessions

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo A Andraus, Principal Investigator — Universidade Norte do Paraná
Locations (1):
- Rodrigo Antonio Carvalho Andraus, Londrina, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hexsel DM, Dal'forno T, Hexsel CL. A validated photonumeric cellulite severity scale. J Eur Acad Dermatol Venereol. 2009 May;23(5):523-8. doi: 10.1111/j.1468-3083.2009.03101.x. Epub 2009 Feb 13. PMID 19220646
- [Result] Yoo MA, Seo YK, Ryu JH, Back JH, Koh JS. A validation study to find highly correlated parameters with visual assessment for clinical evaluation of cosmetic anti-cellulite products. Skin Res Technol. 2014 May;20(2):200-7. doi: 10.1111/srt.12106. Epub 2013 Sep 7. PMID 24010809